CLINICAL TRIAL: NCT03647410
Title: Lumbopelvic Fixation Versus Novel Adjustable Plate for Displaced Sacral Fractures: A Retrospective Cohort Study
Brief Title: Lumbopelvic Fixation Versus Novel Adjustable Plate for Displaced Sacral Fracture
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hebei Medical University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RPZ2018
Record Dates: First submitted 2018-08-21; First posted 2018-08-27 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-06

CONDITIONS: Reduction Deformity of Limb
MeSH Terms: conditions — Ectromelia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lumbopelvic fixation: sacral fractures fixed with lumbopelvic fixation
- novel adjustable plate: sacral fractures fixed with novel adjustable plate
  Interventions: Device: lumbopelvic fixation

INTERVENTIONS:
Device: lumbopelvic fixation — Sacral fractures fixed with lumbopelvic fixation or novel adjustable plate were divided into two groups. Surgical time, intraoperative blood loss, frequency of intraoperative fluoroscopy, reduction quality, related complications, and functional outcome were reviewed.
  Other Names: novel adjustable plate
  Groups: novel adjustable plate

SUMMARY:
Patients of unilaterally displaced sacral fractures fixed with lumbopelvic technique or novel adjustable plate from June 2011 to June 2017 were recruited into this study and were divided into two groups: group A (lumbopelvic fixation) and groups B (novel adjustable plate). Surgical time, intraoperative blood loss, frequency of intraoperative fluoroscopy, reduction quality, related complications were reviewed. Fracture healing was assessed by the radiographs conducted at follow-up. Functional outcome was evaluated according to the Majeed score at the final follow-up.

DETAILED DESCRIPTION:
Patients of unilateral displaced sacral fractures from June 2011 to June 2017 were recruited into this study. The inclusion criteria were as follows: 18-65 years, with normal activity ability before injury, fixed with lumbopelvic technique or novel adjustable plate, completed more than a year follow-up. The exclusion criteria were as follows: pathologic fractures, open fractures, associated with other severe injuries (traumatic brain injury), risk factors affecting bone healing (osteoporosis, smoking, and metabolic diseases) and non-completion of one-year follow-up. Surgical time, intraoperative blood loss, frequency of intraoperative fluoroscopy, related complications were reviewed. Reduction quality was assessed on the postoperative radiographs and CT scans. Functional outcome was evaluated according to the Majeed score system at the final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years, with normal activity ability before injury
* Fixed with lumbopelvic technique or novel adjustable plate
* Completed more than a year follow-up

Exclusion Criteria:

* Pathologic fractures
* Open fractures
* Associated with other severe injuries (traumatic brain injury)
* Risk factors affecting bone healing (osteoporosis, smoking, and metabolic diseases)
* Non-completion of one-year follow-up

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of unilateral displaced sacral fractures from June 2011 to June 2017 were recruited into this study. The inclusion criteria were as follows: 18-65 years, with normal activity ability before injury, fixed with lumbopelvic technique or novel adjustable plate, completed more than a year follow-up. The exclusion criteria were as follows: pathologic fractures, open fractures, associated with other severe injuries (traumatic brain injury), risk factors affecting bone healing (osteoporosis, smoking, and metabolic diseases) and non-completion of one-year follow-up.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-06 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
postoperative reduction quality of sacral fractures after different surgical techniques | 1 year
  maximum displacement distance of the sacral fracture in the postoperative CT scans

SECONDARY OUTCOMES:
the incidence of complication | 1 year
  the incidence of wound infection, iatrogenic injury of vessels and nerves, nonunion

CONTACTS AND LOCATIONS:
Overall Officials: Ruipeng Zhang, Principal Investigator — Third Hospital of Hebei Medical University Department of Orthopaedic Surgery
Locations (1):
- Hebei Medical University Third Hospital, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No